CLINICAL TRIAL: NCT05757349
Title: A Prospective Study on the Prognosis of the Idiopathic Macular Hole With Different Prone Position Times Assisted by Novel Positioning Sensor
Brief Title: Analysis of Novel Positioning Sensor-assisted Postoperative Position Correction and Effective Prone Time Recorded in Patients With Different Prone Times After Macular Hole Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Eye Hospital (Other)
Responsible Party: Principal Investigator, Bojie Hu, Professor, Tianjin Medical University Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TianjinMUEHhbj456
Record Dates: First submitted 2023-02-14; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Idiopathic Macular Hole; Effective Prone Time

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-down position time 1-day group (Experimental): Postoperative face-down position of subjects wearing the novel positioning sensor device for 1-day.
  Interventions: Behavioral: Face-down position time 1-day
- Face-down position time 3-day group (Active Comparator): Postoperative face-down position of subjects wearing the novel positioning sensor device for 3-day.
  Interventions: Behavioral: Face-down position time 3-day

INTERVENTIONS:
Behavioral: Face-down position time 1-day — Postoperative face-down position of subjects wearing the novel positioning sensor device for 1-day.
  Arms: Face-down position time 1-day group
Behavioral: Face-down position time 3-day — Postoperative face-down position of subjects wearing the novel positioning sensor device for 3-day.
  Arms: Face-down position time 3-day group

SUMMARY:
Idiopathic macular hole (IMH) is a fundus disease without clear etiology, most often seen in healthy women over 50 years of age, and is often associated with ocular manifestations such as loss of central vision and visual distortion. It is often associated with loss of central vision, visual distortion, and other ocular manifestations. It is currently treated by vitrectomy combined with internal limiting membranes (ILM) peeling followed by gas filling. A strict prone position for a certain period of time after surgery has a positive effect on the healing of the macular fissure. The need for a strict prone position after IMH has been demonstrated in previous studies (especially when the IMH diameter is >400 μm). However, due to the anti-human mechanics of the face-down position, patient comfort, sleep quality and quality of life are greatly compromised. Therefore, this study designed a smart head position monitoring device to assist patients in maintaining the correct position and recording the effective position time. The study was conducted to determine the shortest prone position time based on macular fissure closure, to minimize the adverse effects of postoperative position, and to obtain the maximum recovery of visual acuity and visual field.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older；
* Patients diagnosed with IMH;
* Patients requiring face-down position after vitrectomy combined with ILM peeling and C3F8(14%) gas filling; Tolerated face-down position after surgery;
* Agreed to the study protocol.

Exclusion Criteria:

* Myopia greater than or equal to -6.0 D; Eye axis length (AL) greater than 26.0mm;
* Trauma, macular edema, macular degeneration, and other secondary MH with clear etiology;
* Previous history of internal eye surgery in the operated eye;
* Patients with local or systemic other diseases significantly affecting visual function;
* Those who cannot maintain face-down position after surgery due to systemic factors, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Macular hole closure rate | 6 month postoperatively
  Ratio of patients with postoperative lacunae that remained closed until the end of the follow-up time to the number of patients who reopened during the follow-up time of those who did not close after surgery
Effective face-down position time | 1 or 3 day postoperatively
  Novel positioning sensor related data cloud storage platform can record and extract effective face-down position time.

SECONDARY OUTCOMES:
Best corrected visual acuity change (BCVA) | 1, 3, 6 month postoperatively
  BCVA for patients after macular fissure surgery, expressed using the (ETDRS) Alphabet Chart.
Retinal nerve fiber layer thickness change | 1, 3, 6 month postoperatively
  Three-dimensional spectral domain optical coherence tomography (SD-OCT)
Macular ganglion cell complex thickness change (GCL+, GCL++) | 1, 3, 6 month postoperatively
  Three-dimensional spectral domain optical coherence tomography (SD-OCT)
Mean retinal Sensitivity (MS) | 1, 3, 6 month postoperatively
  Micro Perimeter 3
Central 2˚ and 4˚ fixation | 1, 3, 6 month postoperatively
  Micro Perimeter 3

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin medical university eye hosipital, Tianjin, Tianjin Municipality, China